CLINICAL TRIAL: NCT03346772
Title: Study of Immune Responses to Influenza Vaccination
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 820590
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Influenza Vaccination
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Influenza vaccination cohort (Experimental): Adults will receive one intramuscular dose of seasonal quadrivalent inactivated influenza vaccine, as indicated for standard of care.
  Interventions: Biological: Influenza vaccination

INTERVENTIONS:
Biological: Influenza vaccination — Adults will receive one intramuscular dose of seasonal quadrivalent inactivated influenza vaccine, as indicated for standard of care.

SUMMARY:
Better understanding of the immune responses to influenza vaccination is needed in order to understand situations of poor vaccine response. Adults will receive influenza vaccination and then have peripheral blood drawn at pre-defined intervals in order to study the lymphocyte responses.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults able to provide consent who need influenza vaccination for standard of care

Exclusion Criteria:

* febrile illness at time of vaccination
* active malignancy
* use of immunosuppressing medications
* blood donation in the past 60 days
* influenza vaccinated during the preceding 6 months
* allergic reactions to influenza vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Influenza neutralizing antibody titers | 21-42 days

CONTACTS AND LOCATIONS:
Overall Officials: E.John Wherry, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No